CLINICAL TRIAL: NCT00720603
Title: Expanded Acess Study of Plerixafor and G-CSF for the Mobilization and Collection of Peripheral Blood Stem Cells for Autologous Stem Cell Transplantation in Patients With Non-Hodgkin's Lymphoma, Hodgkin's Disease or Multiple Myeloma
Brief Title: This is a Multi-center, Single Arm, Open Label Study Intended to Provide Expanded Access to Plerixafor for Patients With Non-Hodgkin's Lymphoma (NHL), Hodgkin's Disease (HD) or Multiple Myeloma (MM) Who Are to Receive Treatment With an Autologous Peripheral Stem Cell Transplant.
Acronym: EAP
Status: No longer available | Type: Expanded Access
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MOZ00607
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma
Keywords: Autologous Stem Cell Transplant
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — plerixafor

INTERVENTIONS:
Drug: Plerixafor — Subcutaneous injection of 240 mcg/kg on the evening prior to each apheresis session
  Other Names: AMD3100, Mozobil

SUMMARY:
The purpose of this program is to provide expanded access to plerixafor for patients with NHL, HD, or MM who are to receive treatment with an autologous peripheral stem cell transplant.

DETAILED DESCRIPTION:
The Expanded Access Program (EAP)(protocol number MOZ00607) is an open label study intended to provide access to plerixafor for patients with non-Hodgkin's Lymphoma, Hodgkin's Disease, or Multiple Myeloma who are to receive treatment with an autologous hematopoietic stem cell transplant. Patients who have previously failed stem cell mobilization attempts or who have previously received an autologous or allogeneic stem cell transplant are not eligible to enroll in this program. The standard of care regimen for stem cell mobilization includes a growth factor, G-CSF, to increase peripheral blood stem cells. Plerixafor is given on the evening prior to doses of standard treatment with G-CSF. The combination of G-CSF and plerixafor has the potential to increase the number of circulating stem cells. The stem cells develop into specialized white blood cells and platelets that are necessary for immune system function and normal blood clotting. The stem cells are removed by a process called apheresis, in which blood is drawn from the patient, the stem cells are separated from the plasma, and the plasma is returned to the patient. The separated stem cells are frozen, similar to the blood banking process. The patient then receives chemotherapy according to the institutional standard. After chemotherapy, stem cell transplant is intended to replenish cells in the bone marrow that may be destroyed by chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM, NHL, or HD.
* Eligible for a planned autologous peripheral stem cell transplantation.
* Written informed consent.
* At least 18 years of age (inclusive).
* Easter Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate cardiac, renal, and pulmonary function sufficient to undergo apheresis and transplantation, I.e., eligible by institutional standards for autologous stem cell transplant.
* Male and female patients of childbearing potential agree to use appropriate form of contraception (i.e., condom, diaphragm cervical cap, etc.) while on study and for at least 3 months following the last treatment. Female patients of child-producing potential must have a negative serum pregnancy test confirmed within 7 days of beginning mobilization therapy.
* White blood cell (WBC) count greater than or equal to 2.5x10^9/L.
* Absolute neutrophil count (ANC) greater than or equal to 1.5x10^9/L.
* Platelet count greater than or equal to 100x10^9/L.
* Serum creatinine less than or equal to 2.2 mg/ dL.
* AST/SGOT, ALT/SGPT, and total bilirubin less than 2.5 x upper limit of normal (ULN).

Exclusion Criteria:

* History of acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), acute myelocytic leukemia (AML), chronic myelocytic leukemia (CML), myelodysplastic syndrome (MDS), plasma cell leukemia or other leukemia.
* Failed previous CD34+ cell collection attempts.
* Prior autologous or allogenic transplantation.
* less than 4 weeks since last anti-cancer therapy (including chemotherapy, biologic/immunologic, radiation) or less than 6 weeks if prior therapy was with nitrosourea or mitomycin (for therapies with prolonged effects, a treatment-free interval of at least 2 half-lives should be considered) with the exception of the following: Treatment with thalidomide, dexamethasone, lenalidomide (Revlimid®), and/or bortezomib (Velcade®) is allowed up to 7 days prior to the first dose of G-CF.
* Bone marrow involvement greater than 20% assessed based on the most recent bone marrow aspirate or biopsy.
* Treated with G-CSF or other cytokine within 14 days prior to the first dose of G-CSF for mobilization.
* HIV positive.
* Active hepatitis B (positive HBsAg) or hepatitis C.
* Acute infection (febrile, i.e., temperature greater than 38 degrees Celsius/100.4 degrees Fahrenheit) within 24 hours prior to dosing or antibiotic therapy within 1 week of enrollment.
* Hypercalcemia as evidenced by greater than 1 mg/dL above ULN.
* Previously received investigational therapy with 4 weeks of enrolling in this protocol or currently enrolled in another investigational protocol during the mobilization phase.
* Central nervous system involvement including brain metastases of leptomeningeal disease.
* Pregnant or nursing women.
* ECG or study result (exercize study, scan) indicative of previously undiagnosed cardiac ischemia or a history of clinically significant rhythm disturbance (arrhythmias), or other conduction abnormality in the last year that in the opinion of the Investigator warrants exclusion of the subject from the trial.
* Co-morbid conditions(s), which in the opinion of the Investigator, renders the patient at high risk from treatment complications or impairs their ability to comply with the study treatment and protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company